CLINICAL TRIAL: NCT01602341
Title: A Multicenter, Randomized, Double-Blind, Four-Week, Bilateral Study of the Safety and Efficacy of Two Concentrations of AN2728 Ointment Administered Once or Twice a Day in Adolescents With Atopic Dermatitis
Brief Title: Efficacy and Safety of AN2728 Topical Ointment to Treat Adolescents With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2728-AD-204
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AN2728 Topical Ointment, 2% QD vs 0.5% QD (Experimental): AN2728 Topical Ointment, 2% applied once daily for 29 days to a target lesion, and AN2728 Topical Ointment, 0.5% applied once daily for 29 days to a target lesion
  Treatments will be randomly assigned to target lesions A and B.
  Interventions: Drug: AN2728 Topical Ointment, 2% QD; Drug: AN2728 Topical Ointment, 0.5% QD
- AN2728 Topical Ointment, 2% BID vs 0.5% BID (Experimental): AN2728 Topical Ointment, 2% applied twice daily for 29 days to a target lesion, and AN2728 Topical Ointment, 0.5% applied twice daily for 29 days to a target lesion.
  Treatments will be randomly assigned to target lesions A and B.
  Interventions: Drug: AN2728 Topical Ointment, 2% BID; Drug: AN2728 Topical Ointment, 0.5% BID

INTERVENTIONS:
Drug: AN2728 Topical Ointment, 2% QD — AN2728 Topical Ointment, 2% QD
  Arms: AN2728 Topical Ointment, 2% QD vs 0.5% QD
Drug: AN2728 Topical Ointment, 0.5% QD — AN2728 Topical Ointment, 0.5% QD
  Arms: AN2728 Topical Ointment, 2% QD vs 0.5% QD
Drug: AN2728 Topical Ointment, 2% BID — AN2728 Topical Ointment, 2% BID
  Arms: AN2728 Topical Ointment, 2% BID vs 0.5% BID
Drug: AN2728 Topical Ointment, 0.5% BID — AN2728 Topical Ointment, 0.5% BID
  Arms: AN2728 Topical Ointment, 2% BID vs 0.5% BID

SUMMARY:
The purpose of this study is to determine the safety and efficacy of AN2728 Topical Ointment, 2% and 0.5%, administered once a day (QD) or twice a day (BID), in the treatment of adolescents with atopic dermatitis (AD)

ELIGIBILITY:
Inclusion Criteria:

* Male or female 12 to 17 years of age, inclusive
* Clinical diagnosis of atopic dermatitis (according to the criteria of Hanifin and Rajka)
* Total body surface area (BSA) of atopic dermatitis involvement ≤35%
* Presence of two comparable target lesions
* Willing and able to comply with study instructions and commit to attending all visits
* Females of childbearing potential must use a highly effective method of birth control. Males with partners of childbearing potential should inform them of their participation in this clinical study and use a highly effective method of birth control during the study.
* Parent/guardian has the ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol-related procedures; subject has the ability to give assent

Exclusion Criteria:

* Significant confounding conditions as assessed by study doctor
* Unstable or actively infected AD
* Active or potentially recurrent dermatologic condition other than atopic dermatitis in the target lesion area that may confound evaluation
* History or evidence of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis)
* Concurrent or recent use of certain topical or systemic medications or phototherapy without a sufficient washout period
* Treatment for any type of cancer (except squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ of the skin, curatively treated with cryosurgery or surgical excision only) within the last 5 years
* Current pregnancy or lactation, or intent to become pregnant during the study
* Known sensitivity to any of the components of the study drug
* Participated in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* Participated in a previous AN2728 clinical study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (11):
  - Anacor Investigational Site, Fremont, California
  - Anacor Investigational Site, Miami, Florida
  - Anacor Investigational Site, Lousiville, Kentucky
  - Anacor Investigational Site, Detroit, Michigan
  - Anacor Investigational Site, Albuquerque, New Mexico
  - Anacor Investigational Site, Stony Brook, New York
  - Anacor Investigational Site, High Point, North Carolina
  - Anacor Investigational Site, Portland, Oregon
  - Anacor Investigational Site, Knoxville, Tennessee
  - Anacor Investigational Site, Salt Lake City, Utah
  - Anacor Investigational Site, Norfolk, Virginia
- Australia (6):
  - Anacor Investigational Site, Phillip, Australian Capital Territory
  - Anacor Investigational Site, Kogarah, New South Wales
  - Anacor Investigational Site, Wooloongabba, Queensland
  - Anacor Investigational Site, Box Hill, Victoria
  - Anacor Investigational Site, Parkville, Victoria
  - Anacor Investigational Site, Fremantle, Western Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily: AN2728 topical ointment, 0.5 percent and 2 percent was applied to 2 anatomically distinct treatment-targeted lesions within each participant with mild to moderate atopic dermatitis (AD), once daily from Day 1 up to Day 29. Lesions were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily: AN2728 topical ointment, 0.5 percent and 2 percent was applied to 2 anatomically distinct treatment-targeted lesions within each participant with mild to moderate AD, twice daily from Day 1 up to Day 28 and applied only once on Day 29. Lesions were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Started | 44 | 42
Completed | 44 | 41
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized and received study drug.
Groups:
- AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily: AN2728 topical ointment, 0.5 percent and 2 percent was applied to 2 anatomically distinct treatment-targeted lesions within each participant with mild to moderate AD, once daily from Day 1 up to Day 29. Lesions were identified at Baseline (Day 1) by investigator.
- Total: Total of all reporting groups
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 42 | 86
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Improvement From Baseline in Atopic Dermatitis Severity Index (ADSI) Score at Day 8
Description: ADSI was used to assess the severity of atopic dermatitis (AD) based on five subscale scores of erythema, pruritus, exudation, excoriation, and lichenification. The severity of each subscale was measured on a 4-point scale ranging from 0 (none) to 3 (severe), where higher scores indicating more severity. ADSI was calculated as the sum of these 5 subscale scores with a total possible score range of 0 (none) to 15 (most severe) where, higher scores indicating more severity. Improvement from Baseline was calculated as Baseline score minus follow-up score.
Time Frame: Baseline, Day 8
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AN2728 Ointment 0.5 Percent, Once Daily: AN2728 topical ointment, 0.5 percent was applied to 1 anatomically distinct treatment-targeted lesion within each participant with mild to moderate AD, once daily from Day 1 up to Day 29. Lesions were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment 2 Percent, Once Daily: AN2728 topical ointment, 2 percent was applied to 1 anatomically distinct treatment-targeted lesion within each participant with mild to moderate AD, once daily from Day 1 up to Day 29. Lesions were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment 0.5 Percent, Twice Daily: AN2728 topical ointment, 0.5 percent was applied to 1 anatomically distinct treatment-targeted lesion within each participant with mild to moderate AD, twice daily from Day 1 up to Day 28 and applied only once on Day 29. Lesions were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment 2 Percent, Twice Daily: AN2728 topical ointment, 2 percent was applied to 1 anatomically distinct treatment-targeted lesion within each participant with mild to moderate AD, twice daily from Day 1 up to Day 28 and applied only once on Day 29. Lesions were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 Ointment 0.5 Percent, Once Daily | AN2728 Ointment 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent, Twice Daily | AN2728 Ointment 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 44 | 42 | 42
units on a scale
  Baseline | 8.22 (1.891) | 8.02 (1.852) | 8.13 (1.811) | 8.19 (1.811)
  Improvement at Day 8 | 2.80 (2.431) | 3.63 (1.695) | 4.33 (2.208) | 4.81 (1.972)

2. Primary Outcome: Improvement From Baseline in Atopic Dermatitis Severity Index (ADSI) Score at Day 15
Description: as for outcome 1
Time Frame: Baseline, Day 15
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Ointment 0.5 Percent, Once Daily | AN2728 Ointment 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent, Twice Daily | AN2728 Ointment 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 44 | 42 | 42
units on a scale | 4.02 (2.781) | 4.34 (2.394) | 4.51 (2.400) | 5.36 (2.028)

3. Primary Outcome: Improvement From Baseline in Atopic Dermatitis Severity Index (ADSI) Score at Day 22
Description: as for outcome 1
Time Frame: Baseline, Day 22
Population: ITT population included all participants, who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Ointment 0.5 Percent, Once Daily | AN2728 Ointment 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent, Twice Daily | AN2728 Ointment 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 44 | 42 | 42
units on a scale | 3.86 (3.157) | 4.55 (2.551) | 4.70 (2.271) | 5.49 (1.803)

4. Primary Outcome: Improvement From Baseline in Atopic Dermatitis Severity Index (ADSI) Score at Day 29
Description: as for outcome 1
Time Frame: Baseline, Day 29
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Ointment 0.5 Percent, Once Daily | AN2728 Ointment 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent, Twice Daily | AN2728 Ointment 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 44 | 42 | 42
units on a scale | 4.47 (3.185) | 5.07 (2.214) | 5.06 (2.361) | 5.81 (1.714)

5. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to Day 29
Population: Safety population included all participants who were randomized and applied at least 1 confirmed dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 42
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Time Frame: Baseline up to Day 29
Population: Safety population included all participants who were randomized and applied at least 1 confirmed dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 42
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug to the end of study treatment (Day 29), that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to Day 29
Population: Safety population included all participants who were randomized and applied at least 1 confirmed dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 42
Participants
  AEs | 6 | 11
  SAEs | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events By Severity
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed on basis of severity as follows: mild=does not interfere with participant's usual function; moderate=interferes to some extent with participant's usual function; severe=interferes significantly with participant's usual function. Number of participants with mild, moderate and severe treatment-emergent AEs were reported in this outcome measure.
Time Frame: Baseline up to Day 29
Population: Safety population included all participants who were randomized and applied at least 1 confirmed dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 42
Participants
  Mild | 6 | 9
  Moderate | 0 | 2
  Severe | 0 | 0

9. Secondary Outcome: Number of Participants With Local Tolerability Symptoms
Description: Participants who experienced local tolerability symptoms: mild itching or burning/stinging at sites of study drug application were reported in this measure.
Time Frame: Baseline up to Day 29
Population: Safety population included all participants who were randomized and applied at least 1 confirmed dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 42
Participants | 3 | 1

10. Secondary Outcome: Improvement From Baseline in ADSI Component Scores (Erythema, Pruritus, Exudation, Excoriation and Lichenification) at Day 8, 15, 22 and 29
Description: ADSI was used to assess the severity of atopic dermatitis (AD) based on five subscale scores of erythema, pruritus, exudation, excoriation, and lichenification. The severity of each subscale was measured on a 4-point scale ranging from 0 (none) to 3 (severe), where higher scores indicating more severity. ADSI was calculated as the sum of these 5 subscale scores with a total possible score range of 0 (none) to 15 (most severe) where, higher scores indicating more severity. Improvement from baseline was calculated as baseline evaluation minus the follow-up evaluation.
Time Frame: Baseline, Day 8, 15, 22, 29
Population: ITT population included all participants who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Ointment 0.5 Percent, Once Daily | AN2728 Ointment 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent, Twice Daily | AN2728 Ointment 2 Percent, Twice Daily
Number analyzed (Participants) | 44 | 44 | 42 | 42
units on a scale
  Erythema: Baseline | 2.23 (0.314) | 2.14 (0.272) | 2.12 (0.216) | 2.15 (0.259)
  Erythema: Improvement at Day 8 | 0.75 (0.678) | 0.90 (0.596) | 0.93 (0.620) | 1.10 (0.637)
  Erythema: Improvement at Day 15 | 1.06 (0.787) | 1.14 (0.702) | 1.13 (0.716) | 1.36 (0.647)
  Erythema: Improvement at Day 22 | 1.02 (0.835) | 1.17 (0.690) | 1.11 (0.610) | 1.40 (0.627)
  Erythema: Improvement at Day 29 | 1.17 (0.785) | 1.17 (0.646) | 1.26 (0.718) | 1.44 (0.636)
  Excoriation: Baseline | 1.43 (0.818) | 1.41 (0.851) | 1.50 (0.819) | 1.50 (0.819)
  Excoriation: Improvement at Day 8 | 0.49 (0.832) | 0.74 (0.633) | 0.88 (0.739) | 1.02 (0.724)
  Excoriation: Improvement at Day 15 | 0.82 (0.778) | 0.78 (0.831) | 0.86 (0.710) | 1.06 (0.790)
  Excoriation: Improvement at Day 22 | 0.68 (0.922) | 0.88 (0.897) | 0.95 (0.731) | 1.08 (0.803)
  Excoriation: Improvement at Day 29 | 0.82 (0.934) | 1.03 (0.824) | 0.96 (0.727) | 1.17 (0.687)
  Exudation: Baseline | 0.77 (0.694) | 0.75 (0.703) | 0.75 (0.751) | 0.80 (0.773)
  Exudation: Improvement at Day 8 | 0.31 (0.531) | 0.49 (0.586) | 0.48 (0.643) | 0.61 (0.668)
  Exudation: Improvement at Day 15 | 0.40 (0.782) | 0.51 (0.796) | 0.42 (0.732) | 0.54 (0.657)
  Exudation: Improvement at Day 22 | 0.40 (0.825) | 0.49 (0.818) | 0.38 (0.688) | 0.57 (0.630)
  Exudation: Improvement at Day 29 | 0.40 (0.839) | 0.57 (0.752) | 0.42 (0.706) | 0.64 (0.710)
  Lichenification: Baseline | 1.67 (0.715) | 1.58 (0.777) | 1.60 (0.692) | 1.58 (0.723)
  Lichenification: Improvement at Day 8 | 0.44 (0.508) | 0.45 (0.480) | 0.65 (0.535) | 0.60 (0.544)
  Lichenification: Improvement at Day 15 | 0.64 (0.554) | 0.59 (0.622) | 0.70 (0.644) | 0.80 (0.681)
  Lichenification: Improvement at Day 22 | 0.55 (0.627) | 0.63 (0.630) | 0.71 (0.554) | 0.77 (0.646)
  Lichenification: Improvement at Day 29 | 0.74 (0.651) | 0.73 (0.686) | 0.79 (0.750) | 0.86 (0.701)
  Pruritus: Baseline | 2.13 (0.582) | 2.15 (0.625) | 2.17 (0.537) | 2.17 (0.502)
  Pruritus: Improvement at Day 8 | 0.82 (0.941) | 1.05 (0.855) | 1.39 (0.753) | 1.50 (0.812)
  Pruritus: Improvement at Day 15 | 1.11 (0.982) | 1.32 (0.857) | 1.40 (0.835) | 1.62 (0.810)
  Pruritus: Improvement at Day 22 | 1.23 (1.026) | 1.39 (0.862) | 1.55 (0.832) | 1.67 (0.770)
  Pruritus: Improvement at Day 29 | 1.35 (1.108) | 1.57 (0.962) | 1.63 (0.699) | 1.71 (0.616)

ADVERSE EVENTS:
Arm/Group | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 6/44 | 11/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AN2728 Ointment 0.5 Percent + 2 Percent, Once Daily (N=44) | AN2728 Ointment 0.5 Percent + 2 Percent, Twice Daily (N=42)
Application site pain (General disorders) | 2 (2) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.